CLINICAL TRIAL: NCT02999412
Title: Medication Reviews Bridging Healthcare: a Cluster-randomised Crossover Trial to Study the Effects of Hospital-initiated Comprehensive Medication Reviews, Including Active Follow-up, on Elderly Patients' Healthcare Utilisation
Brief Title: Medication Reviews Bridging Healthcare: a Cluster-randomised Crossover Trial
Acronym: MedBridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala County Council, Sweden (Other Government)
Collaborators: Region Gävleborg (Other); Västmanland County Council, Sweden (Other Government); Uppsala University (Other); Uppsala Clinical Research Center, Sweden (Unknown)
Responsible Party: Principal Investigator, Thomas Kempen, Principal Investigator, Uppsala County Council, Sweden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: MEDBRIDGE
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Medication Review
Keywords: Integrated Healthcare System; Inappropriate Prescribing; Pragmatic Clinical Trial; Crossover Design; Randomised Controlled Trial
MeSH Terms: interventions — imidazoline I1 receptors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comprehensive medication review (I1) (Active Comparator)
  Interventions: Procedure: Comprehensive medication review
- Comprehensive medication review with active follow-up (I2) (Active Comparator)
  Interventions: Procedure: Comprehensive medication review with active follow-up
- Usual care (Control) (Other)
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Comprehensive medication review — * A thorough medication reconciliation, including a patient/carer interview, by a clinical pharmacist.
  * The clinical pharmacist performs a comprehensive medication review in collaboration with the ward physician and patient, similar to a level three clinical medication review as earlier described in the literature [4]. This includes a structured, critical examination of all of the patient's medications in relation to the patient's conditions, based on information from the patient and the medical record. The objective is to optimise the impact of medications and minimizing the number of medication-related problems. The effects of medication changes will be monitored during the hospital stay by the physician or pharmacist, depending on the specific situation.
  * Before discharge, the clinical pharmacist performs another medication reconciliation to check if the patient's prescriptions for medications to be used after hospital stay are consistent with the patient's medical record.
  Other Names: Intervention 1 (I1)
  Arms: Comprehensive medication review (I1)
Procedure: Comprehensive medication review with active follow-up — The same as I1 but with the following additions:
  * In case of any monitoring needs or necessary subsequent actions to be taken after hospital discharge, the clinical pharmacist and the ward physician send an electronic medication review referral to the patient's primary care physician upon discharge.
  * A first phone call to the patient or carer is made by the clinical pharmacist 2-7 days after the patient is discharged depending on health condition and the pharmacist's availability. This phone call aims to ensure that all information has been understood correctly and to find out if any problems, concerns or questions have arisen after discharge.
  * A second phone call will be made by the clinical pharmacist approximately 30 days after hospital discharge. This phone call aims to find out how the patient is managing the medication and if any problems, concerns or questions have arisen, and to provide the patient with a motivational "boost".
  Other Names: Intervention 2 (I2)
  Arms: Comprehensive medication review with active follow-up (I2)
Procedure: Usual Care — The control group will receive usual hospital care. According to Swedish legislation, usual care includes medication reconciliation upon admission. Next to that, the law requires a medication report addressing the patient's medication treatment to be given to the patient or carer upon hospital discharge and to be attached to the electronic discharge letter. This report contains a motivation and explanation to the changes in medication treatment that have been made during hospital stay, as well as the patient's updated medication list. These mandatory activities are currently carried out to various degree within the different hospitals and wards. Other activities as described in the interventions above may be carried out to a certain degree as well, but no clinical pharmacist will be involved.
  Other Names: Control
  Arms: Usual care (Control)

SUMMARY:
Background: Mismanaged prescribing and use of medication among elderly puts major pressure on current healthcare systems. Performing a medication review, a structured critical examination of a patient's medications, during hospital stay with active follow-up into primary care could optimise treatment benefit and minimise harm. However, a lack of high quality evidence inhibits widespread implementation. This manuscript describes the rationale and design of a pragmatic cluster-randomised, crossover trial to fulfil this need for evidence.

Aim: To study the effects of hospital-initiated comprehensive medication reviews, including active follow-up, on elderly patients' healthcare utilisation compared to 1) usual care and 2) solely hospital based reviews.

Design: Multicentre, three-treatment, replicated, cluster-randomised, crossover trial.

Setting: 8 wards with a multidisciplinary team within 4 hospitals in 3 Swedish counties.

Participants: Patients aged 65 years or older, admitted to one of the study wards. Exclusion criteria: Palliative stage; residing in other than the hospital's county; medication review within the last 30 days; one-day admission.

Interventions: 1, comprehensive medication review during hospital stay; 2, same as 1 with the addition of active follow-up into primary care; 3, usual care.

Primary outcome measure: Incidence of unplanned hospital visits during a 12-month follow-up period.

Data collection and analyses: Extraction and collection from the counties' medical record system into a GCP compliant electronic data capture system. Intention-to-treat-analyses using log-linear Poisson generalized linear mixed models and frailty models.

Relevance: This study has a high potential to show a reduction in elderly patients' morbidity, contributing to more sustainable healthcare in the long run.

DETAILED DESCRIPTION:
Background:

Mismanaged use of multiple medications is one of the greatest risks for healthcare-related harm in the elderly and puts major pressure on current healthcare systems [1,2]. Identifying effective interventions to optimise treatment benefit and minimise harm is an international public health priority [3]. Comprehensive medication review, a structured and critical examination of an individual patient's medications in relation to the patient's conditions, aims to accomplish these goals [4]. A recently published Cochrane meta-analysis examined whether medication reviews lead to improvement in health outcomes of hospitalised adult patients compared with standard care [5]. Ten randomised controlled trials (RCTs) were eventually used for analysis. The authors stated that they "found no evidence that medication review reduces mortality or hospital readmissions, although we did find evidence that medication review may reduce emergency department contacts."[5] A beneficial or detrimental effect on mortality or hospital admissions could be ruled out because estimates were uncertain and follow-up was short. The authors stated that there is a strong need for RCTs of high quality with at least one year follow-up and which are randomised at a cluster level to minimise contamination bias [5]. In addition, a cluster randomised crossover design in which each cluster serves as its own control would increase statistical power [6].

One of the included RCTs in this meta-analysis was conducted by our research group at Uppsala University Hospital in 2005-2006 [7]. We demonstrated in this study that patients, aged 80 years or older, who received a comprehensive medication review including follow-up after hospital discharge, performed by ward based clinical pharmacist, had 16% fewer hospital revisits in the following year. The costs of hospital based care were approximately €200 lower per patient in the intervention group compared to the control group after the intervention costs had been included. The study was conducted on two internal medicine wards with 400 enrolled patients, all 80 years or older, which limits the generalisability of its results.

Today, ten years after our previous RCT, several counties in Sweden have employed clinical pharmacists who perform medication reviews in hospital settings. However, their way of working has changed over time. For this reason it is important to identify the activities that generate the greatest benefits to the patients, which can be done by performing a pragmatic clinical trial, specifically designed to show the real-world effects of such interventions [8]. Therefore we propose this pragmatic cluster-randomised, three-treatment, crossover trial to study the effects of multidisciplinary medication reviews with active follow-up after hospital discharge on elderly patients' healthcare utilisation, compared with solely hospital based reviews and usual care. This large study will generate more robust results and high external validity, with the potential to show effects on hard outcomes such as healthcare utilisation. A similar study has, to our knowledge, not been undertaken anywhere else in the world.

Aim:

To study the effects of hospital-initiated comprehensive medication reviews, including active follow-up, on elderly patients' healthcare utilisation compared to 1) usual care and 2) solely hospital based reviews.

Primary objectives:

1. The first primary objective is to test the hypothesis that the incidence of unplanned hospital visits (admissions plus visits to the emergency department) among elderly patients during a one year follow-up is lower, if they receive a comprehensive medication review with active follow-up after discharge, than if they receive usual care.
2. The second primary objective is to test the hypothesis that a comprehensive medication review with active follow-up after discharge reduces the incidence of unplanned hospital visits more than only a medication review during hospital stay compared to usual care.

Methods:

This study protocol has been developed by using the applicable recommendations of the SPIRIT 2013 Guidance for protocols of clinical trials, the Consort 2010 extension to cluster randomised trials and the Consort 2010 extension to randomized trials of non-pharmacologic treatment [9-11]. The full study protocol is attached to this trial registration.

Setting and clusters:

The study will be conducted in three counties in Sweden: Västmanland, Uppsala and Gävleborg. Within these counties there will be four hospitals taking part in the study: Uppsala University Hospital and the hospitals of Västerås, Enköping and Gävle. At these hospitals clinical pharmacy, including the performance of medication reviews, is an established practice or is planned to be implemented prior to the study. The intervention components of the study will be performed by the existing workforce at two wards within each hospital. The wards differ in terms of medical specialty: geriatric, internal medicine and stroke. All wards are staffed with a multidisciplinary team consisting of physicians, nurses and clinical pharmacists. The pharmacists have either followed a full-time one year post-graduate programme in clinical pharmacy, in which the performance of medication reviews plays a central role, or have followed undergraduate courses in clinical pharmacy and advanced pharmacotherapy. Next to that, all pharmacists have at least six months working experience with performing medication reviews in a multidisciplinary team. To assess clinical skill performance related to medication reviews, all pharmacists participated in an objective structured clinical examination (OSCE), prior to the start of the study. All pharmacists have also participated in a training day with patient case discussions, to assure common practice across all study sites. Other members of the ward team did not receive additional training.

In total eight wards will be included, with each ward acting as a cluster. The study will be carried out as far as possible identically at the eight wards.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to one of the study wards

Exclusion Criteria:

* Has been subject to a medication review within the last 30 days as stated within their medical record;
* Residing in another than the hospital's county
* Being in a palliative stage as stated in their medical record
* Admitted for only one day

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2637 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence of unplanned hospital visits, extracted from the patients' electronic medical record | 12 months
  Admissions plus visits to the emergency department

SECONDARY OUTCOMES:
Unplanned hospital admissions, extracted from the patients' electronic medical record | 30 days
Unplanned hospital admissions, extracted from the patients' electronic medical record | 3 months
Unplanned hospital admissions, extracted from the patients' electronic medical record | 6 months
Unplanned hospital admissions, extracted from the patients' electronic medical record | 12 months
Emergency department visits, extracted from the patients' electronic medical record | 30 days
Emergency department visits, extracted from the patients' electronic medical record | 3 months
Emergency department visits, extracted from the patients' electronic medical record | 6 months
Emergency department visits, extracted from the patients' electronic medical record | 12 months
Unplanned hospital visits, extracted from the patients' electronic medical record | 30 days
  Admissions plus visits to the emergency department
Unplanned hospital visits, extracted from the patients' electronic medical record | 3 months
  Admissions plus visits to the emergency department
Unplanned hospital visits, extracted from the patients' electronic medical record | 6 months
  Admissions plus visits to the emergency department
Unplanned medication-related hospital admissions, extracted from the patients' electronic medical record | 30 days
  Two experienced clinicians will independently assess to what extent the hospital visits were medication-related using the WHO criteria for causality (certain, probable, possible and unlikely). This causality assessment will be based on Case Report Form (CRF) data in which treatment allocation has been blinded, and make use of validated algorithms such as the Naranjo algorithm and the Liverpool ADR Causality Assessment Tool. For a visit to be classified as medication-related consensus needs to be reached between the two clinicians, and where this is not possible, a third expert will have the deciding vote.
Unplanned medication-related hospital admissions, extracted from the patients' electronic medical record | 3 months
  Two experienced clinicians will independently assess to what extent the hospital visits were medication-related using the WHO criteria for causality (certain, probable, possible and unlikely). This causality assessment will be based on Case Report Form (CRF) data in which treatment allocation has been blinded, and make use of validated algorithms such as the Naranjo algorithm and the Liverpool ADR Causality Assessment Tool. For a visit to be classified as medication-related consensus needs to be reached between the two clinicians, and where this is not possible, a third expert will have the deciding vote.
Unplanned medication-related hospital admissions, extracted from the patients' electronic medical record | 6 months
  Two experienced clinicians will independently assess to what extent the hospital visits were medication-related using the WHO criteria for causality (certain, probable, possible and unlikely). This causality assessment will be based on Case Report Form (CRF) data in which treatment allocation has been blinded, and make use of validated algorithms such as the Naranjo algorithm and the Liverpool ADR Causality Assessment Tool. For a visit to be classified as medication-related consensus needs to be reached between the two clinicians, and where this is not possible, a third expert will have the deciding vote.
Unplanned medication-related hospital admissions, extracted from the patients' electronic medical record | 12 months
  Two experienced clinicians will independently assess to what extent the hospital visits were medication-related using the WHO criteria for causality (certain, probable, possible and unlikely). This causality assessment will be based on Case Report Form (CRF) data in which treatment allocation has been blinded, and make use of validated algorithms such as the Naranjo algorithm and the Liverpool ADR Causality Assessment Tool. For a visit to be classified as medication-related consensus needs to be reached between the two clinicians, and where this is not possible, a third expert will have the deciding vote.
Unplanned primary care visits, extracted from the patients' electronic medical record | 30 days
Unplanned primary care visits, extracted from the patients' electronic medical record | 3 months
Unplanned primary care visits, extracted from the patients' electronic medical record | 6 months
Unplanned primary care visits, extracted from the patients' electronic medical record | 12 months
Time from hospital discharge to first unplanned hospital visit, extracted from the patients' electronic medical record | up to 12 months
  time-to-event
Costs of hospital based care, extracted from the counties' costs per patient (CPP) system | 6 months
  Costs for healthcare utilisation including the costs for the intervention. Costs for hospital based healthcare will be retrieved from the counties' CPP system, and average costs for clinical pharmacist employment will be calculated to account for the intervention costs.
Costs of hospital based care, extracted from the counties' costs per patient (CPP) system | 12 months
  Costs for healthcare utilisation including the costs for the intervention. Costs for hospital based healthcare will be retrieved from the counties' CPP system, and average costs for clinical pharmacist employment will be calculated to account for the intervention costs.
All-cause mortality rates, extracted from the national death registry | 30 days
All-cause mortality rates, extracted from the national death registry | 3 months
All-cause mortality rates, extracted from the national death registry | 6 months
All-cause mortality rates, extracted from the national death registry | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Gillespie, Study Chair — Uppsala University Hospital
Locations (4):
- Sweden (4):
  - Gävle Hospital, Gävle, Gävleborg County
  - Enköping Hospital, Enköping, Uppsala County
  - Uppsala University Hospital, Uppsala, Uppsala County
  - Västmanland Hospital, Västerås, Västmanlands Lan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempen TGH, Bertilsson M, Lindner KJ, Sulku J, Nielsen EI, Hogberg A, Vikerfors T, Melhus H, Gillespie U. Medication Reviews Bridging Healthcare (MedBridge): Study protocol for a pragmatic cluster-randomised crossover trial. Contemp Clin Trials. 2017 Oct;61:126-132. doi: 10.1016/j.cct.2017.07.019. Epub 2017 Jul 21. PMID 28739539
- [Background] Kempen TGH, Hedstrom M, Olsson H, Johansson A, Ottosson S, Al-Sammak Y, Gillespie U. Assessment tool for hospital admissions related to medications: development and validation in older patients. Int J Clin Pharm. 2019 Feb;41(1):198-206. doi: 10.1007/s11096-018-0768-8. Epub 2018 Dec 26. PMID 30585296
- [Result] Kempen TGH, Kalvemark A, Gillespie U, Stewart D. Comprehensive medication reviews by ward-based pharmacists in Swedish hospitals: What does the patient have to say? J Eval Clin Pract. 2020 Feb;26(1):149-157. doi: 10.1111/jep.13121. Epub 2019 Mar 4. PMID 30834647
- [Result] Kempen TGH, Cam H, Kalvemark A, Lindner KJ, Melhus H, Nielsen EI, Sulku J, Gillespie U. Intervention fidelity and process outcomes of medication reviews including post-discharge follow-up in older hospitalized patients: Process evaluation of the MedBridge trial. J Clin Pharm Ther. 2020 Oct;45(5):1021-1029. doi: 10.1111/jcpt.13128. Epub 2020 Mar 14. PMID 32171028
- [Result] Kempen TGH, Kalvemark A, Sawires M, Stewart D, Gillespie U. Facilitators and barriers for performing comprehensive medication reviews and follow-up by multiprofessional teams in older hospitalised patients. Eur J Clin Pharmacol. 2020 Jun;76(6):775-784. doi: 10.1007/s00228-020-02846-8. Epub 2020 Feb 19. PMID 32076745
- [Result] Kempen TGH, Bertilsson M, Hadziosmanovic N, Lindner KJ, Melhus H, Nielsen EI, Sulku J, Gillespie U. Effects of Hospital-Based Comprehensive Medication Reviews Including Postdischarge Follow-up on Older Patients' Use of Health Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e216303. doi: 10.1001/jamanetworkopen.2021.6303. PMID 33929523
- See also: Official study website — http://www.akademiska.se/MedBridge

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with summarized SAP (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT02999412/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT02999412/SAP_001.pdf